CLINICAL TRIAL: NCT03959878
Title: Feasibility of a Constant Pressure Skin Disk (CPSD) in Enteral Tubes.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-001922
Record Dates: First submitted 2018-03-20; First posted 2019-05-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gastrostomy
Keywords: Jejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Gastrostomy Tube (Experimental): Non-hospitalized outpatients undergoing placement of a gastrointestinal gastrostomy tube (GIG tube) or GI jejunostomy tube (GIJ tube) will receive the usual Standards of Care related to the placement of a GIG or GIJ tube and the Constant Pressure Skin Disk.
  Interventions: Device: Constant Pressure Skin Disk

INTERVENTIONS:
Device: Constant Pressure Skin Disk — The external disk is made of Dow Corning® Silastic Q7-4850 liquid silicone rubber. Placement of the disk will be done by the gastroenterologist or interventional radiologist during the gastrointestinal gastrostomy tube (GIG) or gastrointestinal jejunostomy tube (GIJ) placement procedure. The gastroenterologist or interventional radiologist will replace the manufacturer's external, adjustable skin disk with the external, adjustable Constant Pressure Skin Disk, by sliding the former off and the latter on to the feeding tube.

SUMMARY:
Researchers are gathering information on one specific part of a feeding tube, known as the adjustable skin disk. Researchers are trying to see if a new type of adjustable skin disk, called a Constant Pressure Skin Disk (CPSD), can safely and effectively support adequate healing, and reduced complication rates.

DETAILED DESCRIPTION:
During the procedure of placing a gastrointestinal gastrostomy tube (GIG tube) or GI jejunostomy tube (GIJ tube), the gastroenterologist or interventional radiologist will replace the manufacturer's external, adjustable skin disk with the external, adjustable Constant Pressure Skin Disk (CPSD) by sliding the former off and the latter on to the feeding tube.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 22 years
* Undergoing PEG tube or PEJ tube placement

Exclusion Criteria:

* History of tobacco or illegal drug use in the past year
* History of an enteral tube
* History of gastric surgery (bariatric surgery, Nissen fundoplication, etc.)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Constant Pressure Skin Disk (CPSD) durability | 180 days
  Number of devices that remain intact

SECONDARY OUTCOMES:
Adverse Events | 180 days
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet S Mundi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials